CLINICAL TRIAL: NCT07256795
Title: Blood-Brain Barrier Integrity and Immune Dynamics in Neuropsychiatric Sequelae of Post-SARS-CoV-2 Onset ME/CFS Versus Pre-Pandemic ME/CFS Patients
Acronym: MECFS BBB
Status: Not yet recruiting | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00537228
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Chronic Fatigue Syndrome
MeSH Terms: conditions — Fatigue Syndrome, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Myalgic Encephalomyelitis/Chronic Fatigue Syndrome (ME/CFS) is a complex chronic illness impacting multiple body systems and characterized by activity-limiting fatigue and post exertional symptom exacerbation, affecting over 3.5 million adults in the US and as many as half of those with long COVID. The mechanisms behind the frequently profound cognitive impairments in MECFS are elusive; however, disruption of the integrity of the blood brain barrier (BBB) and immune cell migration into the brain are thought to contribute to neuroinflammation and related neuropsychiatric burden in MECFS. This project combines brain imaging, neuropsychiatric assessments, and blood-based measures of inflammation in pre-pandemic and post-pandemic individuals with MECFS to understand the role of BBB permeability and inflammation as contributors to key aspects of cognition and mood.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for pre-pandemic onset ME/CFS cohort:
* 18-70 years of age
* At least 8th grade education
* Onset of the following symptoms prior to July 2019 (Pre-SARS-CoV-2 pandemic) and meeting 2015 IOM diagnostic criteria for MECFS:
* Substantial reduction in functioning and persistent and profound fatigue for at least 6 months. The person is unable to undertake the same level of activity before they became - . Their fatigue is not the result of significant exertion and is not substantially alleviated by rest.
* Post-exertional malaise.
* Unrefreshing sleep
* At least one of the following two symptoms:
* Cognitive impairment (difficulty with memory, finding words, understanding etc).
* Orthostatic intolerance (symptoms like palpitations, sweating, dizziness, nausea when standing that are reduced or eliminated when lying down).

Inclusion criteria post SARS-CoV-2 onset ME/CFS:

* 18-70 years of age
* At least 8th grade education
* Previous suspected, probable, or confirmed SARS-CoV-2 infection, as defined by the World Health Organization:
* Suspected case of SARS-CoV-2 infection
* Three options, A through C:

Meets the clinical OR epidemiological criteria.

* Clinical criteria: Acute onset of fever AND cough (influenza-like illness) OR Acute onset of ANY THREE OR MORE of the following signs or symptoms: fever, cough, general, weakness/fatigue, headache, myalgia, sore throat, coryza, dyspnea, nausea, diarrhea, anorexia.
* Epidemiological criteria: Contact of a probable or confirmed case or linked to a COVID-19 cluster; or B. Presents with acute respiratory infection with history of fever or measured fever of ≥ 38°C; and cough; with onset within the last 10 days; and who requires hospitalization) C. Presents with no clinical signs or symptoms, NOR meeting epidemiologic criteria with a positive professional use or self-test SARS-CoV-2 antigen-Rapid Diagnostic Test.
* Probable case of SARS-CoV-2 infection, defined as meets clinical criteria above AND is a contact of a probable or confirmed case or is linked to a COVID-19 cluster.
* Confirmed case of SARS-CoV-2 infection - Two options, i. and ii.:
* A person with a positive nucleic acid amplification test, regardless of clinical criteria OR epidemiological criteria; or
* Meeting clinical criteria AND/OR epidemiological criteria (See suspect case A). With a positive professional use or self-test SARS-CoV-2 Antigen-Rapid Diagnostic Test.
* Post SARS CoV 2 onset of the following symptoms, meeting 2015 IOM diagnostic criteria for ME/CFS:
* Substantial reduction in functioning and persistent and profound fatigue for at least 6 months. The person is unable to undertake the same level of activity before they became - - Their fatigue is not the result of significant exertion and is not substantially alleviated by rest.
* Post-exertional malaise.
* Unrefreshing sleep.
* At least one of the following two symptoms:
* Cognitive impairment (difficulty with memory, finding words, understanding etc).
* Orthostatic intolerance (symptoms like palpitations, sweating, dizziness, nausea when standing that are reduced or eliminated when lying down).
* Given that our application focuses on MECFS patients with neuropsychiatric symptoms the investigators will require participants to report >1 symptom with at least one of the symptoms being neuropsychiatric in nature (e.g., brain fog, anxiety, depression, headaches).

Exclusion both groups (pre-pandemic onset ME/CFS and post SARS-CoV-2 onset ME/CFS):

* History of Axis I psychiatric disorders (including alcohol and drug dependence) except for mood disorders which developed after onset of ME/CFS symptoms.
* Severe or unstable medical condition that would interfere with physical participation.
* Neurological disorders, such as stroke, epilepsy, multiple sclerosis, Parkinson's disease, or dementia.
* History of severe head injury that resulted in persistent traumatic brain injury sequelae.
* Any condition that is contraindicated for the MRI environment (e.g., metal in the body, pacemaker, claustrophobia)
* Currently pregnant.
* Lack of English proficiency (to ensure validity in verbal outcome measures)
* Active or recent (within 3 months) substance misuse (which is known to affect BBB permeability) assessed by clinical interview and toxicology (nicotine/cannabis allowed)
* History of psychosis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 18-70 years of age
  * At least 8th grade education
  * Onset of the following symptoms prior to July 2019 (Pre-SARS-CoV-2 pandemic) and meeting 2015 IOM diagnostic criteria for MECFS:
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2030-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Permeability Surface-Area Product (PS) | Up to 5 years
  Investigate BBB permeability in MECFS patients using WEPCAST MRI as measured by Permeability Surface-Area Product (PS)
Inflammatory biomarkers levels | Up to 5 years
  Inflammatory biomarkers levels and their relation to BBB or and its relationship to cognitive impairments

CONTACTS AND LOCATIONS:
Overall Officials: Alba Azola, MD, Principal Investigator — Johns Hopkins University